CLINICAL TRIAL: NCT05759416
Title: Evaluation of the Efficacy of Topically Applied Melatonin Gel as Adjunctive Therapy in Chronic Periodontitis; Randomized Control Trial
Brief Title: Evaluation Efficacy of Melatonin Gel as Adjunctive Therapy in Chronic Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Shaymaa Hussein Rafat Kotb, principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AADJ-2111-1091; Aadj@azhar.edu.eg (Registry Identifier: ISSN 2682-2822)
Record Dates: First submitted 2023-01-13; First posted 2023-03-08 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis; Melatonin; RANKL (Receptor activator nuclear K ligand); ELISA (Enzyme-Linked Immunosorbent Assay); Gingival crevicular fluid
MeSH Terms: conditions — Chronic Periodontitis; Osteopetrosis, mild autosomal recessive form

STUDY DESIGN:
Intervention Model Description: Forty chronic periodontitis selected patients ,divided into two groups. Group I: included 20 chronic periodontitis patients, treated by conventional periodontal therapy SRP combined with intra- pocket application of Melatonin gel once weekly for 1 month begin application at the second week after initial therapy. Group II: included 20 chronic periodontitis patients, treated by SRP combined with the injection of placebo, weekly for one month.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gp I(Melatonin gp) (Active Comparator): Group I: included 20 chronic periodontitis patients, treated by conventional periodontal therapy SRP combined with intra- pocket application of Melatonin gel once weekly for 1 month begin application at the second week after initial therapy.
  Interventions: Drug: Melatonin2%gel
- Gp II(placebo gp) (Placebo Comparator): Group II: included 20 chronic periodontitis patients, treated by SRP combined with the injection of placebo, weekly for one month
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Melatonin2%gel — Intra-pocket application of 2% Melatonin gel
  Other Names: intra- pocket Melatonin gel
  Arms: Gp I(Melatonin gp)
Drug: PLACEBO — placebo intra-pocket application
  Arms: Gp II(placebo gp)

SUMMARY:
This study was conducted to assess the benefit of locally delivered melatonin gel as adjunctive to scaling and root planning (SRP) in the treatment of chronic periodontitis.

DETAILED DESCRIPTION:
Forty chronic periodontitis selected patients ,divided into two groups. Group I: included 20 chronic periodontitis patients, treated by conventional periodontal therapy SRP combined with intra- pocket application of Melatonin gel once weekly for 1 month begin application at the second week after initial therapy. Group II: included 20 chronic periodontitis patients, treated by SRP combined with the injection of placebo, weekly for one month. The periodontal parameters were recorded at baseline, 1week, 1and 3 months.Gingival crevicular fluid (GCF) samples were collected and a quantitative measurement of receptor activator nuclear K ligand (RANKL) was carried out by using Enzyme-Linked Immunosorbent Assay (ELISA) at baseline, 1week, 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosed with chronic periodontitis , must be able to maintan good oral hygiene

Exclusion Criteria:

Diabetic mellitus immunsuppressive medication

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Melatonin gel by determine the change on measurements of clinical parameter in chronic periodontitis. | 2 weeks
  positive change in clinical parameter by millimeter
EFFICACY of Melatonin Gel by positive change measurements of clinical parameter "pocket depth ,attachment loss" | 1: 3 months
  positive change in clinical parameter by millimeter

SECONDARY OUTCOMES:
EFFICACY of Melatonin Gel by positive change on concentration level of Receptor activator nuclear K ligand ( RANKL) in Gingival crevicular fluid (GCF) | 3 months
  microbiology analysis by Receptor activator nuclear K ligand(ELISA ) by picogram

OTHER OUTCOMES:
pre-opertive measurements of clinical parameter in chronic periodontitis | at beginning of trial
  negative result in clinical parameter measurments by millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar university ,faculty of Dental Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
yes ,no problem to share study result
Supporting Information: Study Protocol, SAP, CSR
Time Frame: any time .It is already published
Access Criteria: DOI: 10.21608/aadj.2022.267325
URL: https://aadj.journals.ekb.eg/article_234723.html

REFERENCES:
- [Result] kotb, shaymaa Hussein Rafat
- See also: shaymaa+kotb@orcid — https://orcid.org/my-orcid?orcid=0000-0002-8404-438X

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT05759416/Prot_SAP_000.pdf